CLINICAL TRIAL: NCT06896474
Title: SDM POSSIBLE: A Cluster RCT of a Breast Cancer Treatment Decision Aid for Women 70+ With Low-Risk Stage I Breast Cancers
Brief Title: SDM POSSIBLE: A Breast Cancer Treatment Decision Aid for Women 70+ With Low-Risk Stage I Breast Cancers
Acronym: SDMPOSSIBLE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Mara Schonberg, Principal Investigator, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 24-565
Record Dates: First submitted 2025-03-18; First posted 2025-03-26 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Breast Neoplasm; Breast Neoplasms; Breast Cancer; ER+ Breast Cancer; HER2-negative Breast Cancer
Keywords: Breast Neoplasm; Breast Neoplasms; Breast Cancer; ER+ Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Decision Support Techniques; SDM

STUDY DESIGN:
Intervention Model Description: Cluster randomized controlled trial at the surgeon level
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Surgeons + SDM/DA (Experimental): 22 enrolled surgeon participants will be randomized and will complete:
  * Baseline questionnaire
  * Virtual 1 hour training on SDM
  * 3-month training follow up survey
  * At Month 12: 6 surgeon participants will take part in a semi-structured interview with research assistant/PI by phone, in-person, or virtually
  * End-of-study survey
  * At end of study 6 surgeon participants will take part in a semi-structured interview with research assistant/PI by phone, in-person, or virtually.
  Approximately, 153 patients and 17 caregivers will be in this arm. They will complete a survey at 1 week and 6 months. At 12 months investigators will ask 12 patients and 4 caregivers to complete a qualitative interview. At end of study investigators will ask 12 patients and 4 caregivers to complete a qualitative semi-structured interview with research assistant/PI by phone, in-person, or virtually.
  Interventions: Behavioral: Shared Decision-Making Training and Decision Aid
- Standard-of-Care (No Intervention): 22 enrolled surgeons will be randomized to usual care and will complete:
  * Baseline questionnaire
  * End-of-study survey
  * May choose to participat in End-of-study virtual 1 hour training on SDM
  * 3-month training follow up survey evaluating the training
  Approximately, 153 patients and 17 care-givers will be in this arm. They will complete a survey at 1 week and 6 months.

INTERVENTIONS:
Behavioral: Shared Decision-Making Training and Decision Aid — The intervention includes training surgeons in shared decision making techniques and providing eligible participants with a tailored breast cancer treatment decision aid prior to the initial surgical consultation.
  Other Names: SDM and DA
  Arms: Surgeons + SDM/DA

SUMMARY:
Investigators aim to conduct a type 1 hybrid effectiveness-implementation surgeon-level cluster randomized clinical trial (RCT) of a multi-level intervention, a shared decision making training for surgeons plus patient decision aid vs. usual care (UC), at 6 large health systems in 4 regions to learn the intervention's effectiveness. Decision aids will be mailed and sent via patient portal and/or via email (when portal/email addresses are available) to patients before their first surgical encounter. The central hypothesis is that the novel intervention will be a key resource to support shared decision making leading to higher quality treatment decisions and as result improved care and outcomes.

DETAILED DESCRIPTION:
In a parallel group-randomized trial, investigators aim to test the effects of training breast surgeons in shared decision making and providing their female patients aged 70 and older with Stage 1 (2 centimeters or less), estrogen receptor positive (ER+), human epidermal growth factor receptor 2 negative (HER2-) breast cancer a patient decision aid on breast cancer treatment. The decision aid is novel in that it includes comprehensive information about the benefits and harms of the different breast cancer treatments that older woman may be offered. It also highlights the complex interplay between their multiple treatment options and their health, life expectancy, values and preferences.

The investigators plan to recruit 44 surgeons from six different health systems (including Beth Israel Lahey Health, Dana Farber Cancer Institute, University of Rochester, Duke University Medical Center, City of Hope, and Rutgers University) to participate in this trial. To participate, a surgeon must agree to complete a previously developed 1-hour training in shared decision making and to allow their eligible patients to be sent the patient decision aid if randomized to the intervention. In order to participate, surgeons must also complete a baseline survey that takes <2 minutes to complete and asks surgeons 6 questions about how confident they are in engaging older women in shared decision making around breast cancer treatment. Surgeons must confirm that they consent to participate on the baseline survey.

Once a surgeon agrees to participate and completes the baseline survey they will be randomized to either the intervention arm or to the usual care arm. Surgeons randomized to the usual care arm will continue with their usual treatment discussions without being provided any support for shared decision making so that investigators may learn the effects of the intervention compared to real-world practice. Investigators will wait 8 weeks after a surgeon completes the baseline survey before following eligible patients in their panel to allow surgeons randomized to the intervention arm time to participate in the shared decision making training. Dr. Schonberg, the principal investigator of this study, will offer many times and make herself widely available to intervention arm surgeons to provide the live televideo training in shared decision making. If the 8 week mark is approaching and the intervention arm surgeon has not been able to schedule a time to complete the training, then Dr. Schonberg will send the surgeon a video copy of the training to watch. During the training, surgeons practice shared decision making using their own language. Intervention arm surgeons will also receive access to a secure website with all the decision support tools and strategies discussed in the training. In addition, investigators will invite intervention arm surgeons to submit challenging cases of decision making with women aged 70 and older with Stage I, ER+, HER2- breast cancer for feedback throughout the trial. The research team will send any feedback shared and updates in shared decision making to all intervention arm surgeons throughout the trial through a study newsletter every 6 months. Every year, investigators will thank surgeons in both arms for their participation and will send them an update regarding study recruitment.

To identify patients in participating surgeon panels who may be eligible to receive the decision aid, a research assistant (RA) at each site will review the appointment logs of participating surgeons at least twice a week during the trial to identify eligible women. Women aged 70 and older with Stage I, ER+, HER2- breast cancer are eligible to receive the decision aid if they are English or Spanish-speaking since the decision aid has been developed in English and Spanish. RAs will mail all patients the decision aid via express mail (or overnight mail if needed to reach the patient before their first surgical encounter). RAs will also email patients the decision aid if they have an email listed in the electronic medical record (EMR) and they will send the decision aid to patients via the patient portal if the patient has registered with the portal. When sending patients the decision aid, RAs will include a cover letter that explains the purpose of the decision aid (that it was designed to support communication between breast surgeons and women age 70 and older) and that some women may find it helpful to read the decision aid before, during, or right after their first visit with their breast surgeon.

To learn the effect of the intervention on treatments received by women aged 70 and older with Stage I, ER+, HER2- breast cancer, a RA will review the medical records of all patients with eligible tumor and study characteristics in a participating surgeon's panel to see what treatments they received within six months of their initial surgical visit. The chart abstraction instrument assesses whether a patient received a mastectomy, lumpectomy, radiation therapy, lymph node surgery, and endocrine therapy as well as any comorbidities listed in the patient's problem list. At the end of the study, the research assistant will also review patients' medical records to learn if the patient experienced a breast cancer recurrence, is still alive, and if not, the cause of death. Investigators will follow patients for this information between 6 months and 3.5 years depending on when the patient is seen by a participating surgeon during the trial.

To better understand variation in surgeon treatment patterns at baseline, investigators will also conduct a retrospective chart review to review treatments received by women aged 70 and older with clinically node-negative, <2cm, ER+, HER2- breast cancer within one year prior to a surgeon's completing the study's baseline surgeon questionnaire to learn their baseline likelihood to treat women >70, English/Spanish speaking, diagnosed with a first primary <2cm, clinically node negative, ER+, HER2- breast cancer with mastectomy, Sentinel lymph node biopsy (SLNB), or RT after BCS.

Investigators will also ask all surgeons to complete a brief end-of-study survey (<5 minutes to complete) that asks surgeons again the 6 questions about how confident they are in engaging older women in shared decision making around breast cancer treatment and their attitudes towards shared decision making around breast cancer treatment with older women. Surgeons will also be asked to share their thoughts on the decision aid. Since the trial will be complete, the survey will include a link to the decision aid that surgeons in both arms may review to provide feedback on the decision aid. After completing the end-of-study survey, investigators will invite surgeons randomized to the usual care arm to participate in the shared decision making training. All surgeons who participate in the training will be asked to complete an evaluation of the training 6 months later. This time period will allow surgeons time to practice what they learn in the training before completing the evaluation survey. Surgeons randomized to the intervention arm will complete this evaluation 6 months after being trained in shared decision making during the trial while surgeons randomized to the usual care arm will complete this evaluation at least 6 months after the trial has ended since these surgeons can only be trained in shared decision making after the trial has ended. Investigators anticipate surgeons will complete study surveys via a secure web-link; however, investigators will offer surgeons to have a research assistant administer the survey to them or to complete a paper copy of the survey if they prefer.

Investigators aim to recruit at least 44 surgeons practicing at recruitment sites. They further anticipate that these 44 surgeons will see at least 1,120 women eligible to receive the decision aid during the three years of the trial (~25 patients overall or 8-9 women per year per surgeon). With these numbers investigators anticipate being able to show that 15% fewer patients seen by an intervention arm surgeon will receive low-value care including a mastectomy, radiation after breast conserving surgery or a lymph node biopsy compared to patients who receive care from a usual care arm surgeon, assessed administratively.

Investigators also anticipate that at least 32 surgeons will complete both a baseline study questionnaire and an end-of-study questionnaire which will allow the investigators to detect if there is about a 1-point improvement in the 6-item index evaluating surgeon self-confidence to engage older women in shared decision making around breast cancer treatment (each item is scored 1-7 points and the total score is determined by calculating the mean score on the 6-item index).

In Aim 2, investigators aim to recruit a subset of patients seen by surgeons participating in the Aim 1 parallel group-randomized trial to complete study surveys to capture participant reported outcomes about the intervention (which includes training breast surgeons in shared decision making and providing women aged 70 and older with Stage I [2 centimeters of less], ER+, HER2- breast cancers with a patient decision aid.) Investigators aim to recruit 340 patients or caregivers for women who would not be able to participate because of memory loss to complete a study survey approximately one week after their first surgical encounter and six months later. The investigators estimate that 34 patients will have a caregiver complete the study surveys and they anticipate that 306 women will complete study surveys for themselves. A research assistant will attempt to approach eligible patients seen by a participating surgeon at the time of their initial surgical visit to ask them if they are willing to participate. English and Spanish speaking females without a prior history of breast cancer who have been newly diagnosed with a Stage I [2 centimeters of less], ER+, HER2- breast cancer are eligible since the decision aid being tested was developed for these patients. Investigators do not plan to include biological males since the data informing the decision aid were obtained from studies of biological females and treatment recommendations and outcomes tend to be worse for biological males with breast cancer.

For patients/caregivers who agree to participate, a research assistant (RA) will offer to administer the 1-week survey in person after the visit, to administer the 1-week survey over the telephone in the next three weeks as long as the patient has not yet undergone surgery at the time of the 1-week survey, or to send the patient/caregiver a secure web-link or a paper copy (based on patient/caregiver preference) for the patient/caregiver to self-administer the survey.

The 1-week survey asks patients/caregivers about the quality of shared decision making with their surgeons, their knowledge of the benefits and harms of different breast cancer treatments, their decisional conflict around treatment, their health related quality of life, their preferred role in treatment decisions, their perceived involvement in treatment decisions, and where they are at in terms of treatment decision making. It also asks patients/caregivers their sociodemographics. The 6-month survey asks patients/caregivers about the quality of shared decision making with their radiation oncologists and oncologists, their knowledge of the benefits and harms of endocrine therapy, their decisional conflict around treatment, their health related quality of life, the financial burden of treatment, their satisfaction with their treatment decisions, whether they have any regret about the decisions made, their perceived involvement in treatment decisions, which treatments they received, and about their health care utilization. For patients/caregivers whose surgeon is randomized to the intervention arm, investigators will ask them about their use of the decision aid, whether it was acceptable to them, and whether it prepared them for decision-making. RAs will offer to administer the 6-month survey in person, over the telephone, or to send the patient/caregiver a secure web-link to the survey or a paper copy (based on patient/caregiver preference) for the patient/caregiver to self-administer the survey.

Finally, investigators will use information that patients/caregivers provide on treatments received, health care utilization, and time spent reviewing/delivering the decision aid and training surgeons in shared decision making to determine the costs of our intervention and the costs of care for patients in the usual care arm compared to those in the intervention arm. Investigators will also examine whether there are differences by arm in patient/caregiver health related quality of life. If healthcare costs of patients in the intervention arm are less than those in the usual care arm and their quality of life is better it will be clear that the intervention is a high quality and low cost intervention. If healthcare costs of patients in the intervention arm are higher than those in the usual care arm but their quality of life is better investigators will examine the cost threshold for improved quality life of patients.

In Aim 4, investigators will conduct semi-structured individual qualitative interviews with intervention arm patients (n=12), and caregivers (n=4) and intervention arm surgeons (n=6) at 12 months to learn their thoughts on how implementation of the intervention has gone. At the end-of-study, investigators will also conduct semi-structured individual qualitative interviews with intervention arm patients (n=12), and caregivers (n=4) and intervention arm surgeons (n=6) to learn how best to implement and disseminate the intervention. At the end of the study, investigators will also interview at least 6 administrators and 12 allied health professionals referred by intervention arm surgeons to learn their perspectives on how best to implement the intervention.

In summary, it is expected about 402 people will participate in this research study including 44 surgeons, 306 women aged 70 and older newly diagnosed with 2cm or less, clinically lymph node negative, estrogen receptor positive, HER2- breast cancer without memory problems, 34 of caregivers of women aged 70 and older newly diagnosed with 2cm or less, clinically lymph node negative, estrogen receptor positive, HER2- breast cancer with memory problems, and 18 administrators and/or allied healthcare professionals.

ELIGIBILITY:
Surgeon Inclusion Criteria:

* Non-resident surgeon >18 years old
* Cares for women >/= 70 years at one of the recruitment practices.
* Ability and willingness to provide verbal consent

Aim 1 Participant Inclusion Criteria: Participants whose medical records will be followed for treatments received and survival

* Biological female
* aged 70 or older
* first primary invasive breast cancer
* clinically </=2 cm
* clinically lymph node negative
* estrogen receptor positive (ER+) -HER2-
* scheduled with a participating surgeon for an initial encounter. Females with ER+ breast cancer will be included regardless of their progesterone receptor (PR) status since treatment decisions are similar for ER+/PR+ and ER+/PR- women.

Aim 1 Participant Inclusion Criteria: Participants whose medical records will be reviewed retrospectively for treatments received in the year before the participating surgeon completes the baseline questionnaire

* Biological female
* aged 70 or older
* a first primary invasive breast cancer
* clinically </=2 cm
* clinically lymph node negative
* estrogen receptor positive(ER+) -HER2-
* saw a participating surgeon for an initial encounter in the year before the surgeon completed the baseline questionnaire.

Aim 2 Participant Inclusion Criteria: Participants who will be included in Aim 2 participant surveys to learn patient reported outcomes

* Biological female
* aged 70 or older
* first primary invasive breast cancer
* clinically </=2 cm
* clinically lymph node negative
* estrogen receptor positive (ER+) -HER2-
* scheduled with a participating surgeon for an initial encounter. If a patient completes the baseline questionnaire and then is found to have different tumor characteristics (e.g., found to be lymph node positive during surgery), investigators plan to retain the patient in the study and ask them to complete the second survey.

Primary caregiver Inclusion Criteria:

* primary family, friend, or non-paid caregiver (herein referred to as caregiver) of a patient unable or unwilling to complete study questionnaires due to cognitive decline. The primary family, friend, or non-paid caregiver will be identified by the patient, self-identified, or documented as the decision maker in the medical record.
* Age >18
* English or Spanish speaking
* Ability and willingness to provide verbal consent

Allied health professionals (Aim 4 at the end of the trial) Inclusion Criteria:

* Administrator, social worker, physician assistant, navigator, nurse or other allied health professional in breast surgery
* Ability and willingness to provide verbal consent

Surgeon Exclusion Criteria:

* Resident surgeon
* Non-surgeons
* Psychiatric illness situations that would limit compliance with study requirements

Aim 1 Participant Exclusion criteria: Participants whose medical records will be followed for treatments received and survival

* Age <70
* Biological males: Biological males will be excluded since the data informing the DA were obtained from studies of biological females and treatment recommendations and outcomes tend to be worse for biological males with breast cancer.
* Non English or non-Spanish speaking: Women who do not speak English or Spanish will be excluded since these women are not eligible for the DA.
* History of invasive breast cancer
* History ductal carcinoma in situ treated with radiation (since these women are generally not be eligible for radiation treatment)
* Women with Paget's disease because treatment options differ
* inflammatory breast cancer because treatment options differ
* Phyllodes tumor because treatment options differ.
* In hospice
* Surgeon not willing to participate

Aim 1 Participant Exclusion Criteria: Participants whose medical records will be reviewed retrospectively for treatments received in the year before the participating surgeon completes the baseline questionnaire

* Age <70
* Biological males: Biological males will be excluded since the data informing the DA were obtained from studies of biological females and treatment recommendations and outcomes tend to be worse for biological males with breast cancer.
* Non English or non-Spanish speaking: Women who do not speak English or Spanish will be excluded since these women are not eligible for the DA. If the DA is found to be effective in English and Spanish we plan to have the DA professionally translated to other languages at the end of the trial. English and Spanish are the most common languages spoken by older women at our recruitment sites.
* History of invasive breast cancer
* History ductal carcinoma in situ treated with radiation (since these women are generally not be eligible for radiation treatment)
* Paget's disease inflammatory breast cancer
* Phyllodes tumor
* In hospice
* Surgeon not willing to participate

Aim 2 Participant Exclusion Criteria: Participants who will be included in Aim 2 participant surveys to learn patient reported outcomes

* Age <70
* Biological males: Biological males will be excluded since the data informing our DA were obtained from studies of biological females and treatment recommendations and outcomes tend to be worse for biological males with breast cancer.
* Non English or non-Spanish speaking: Women who do not speak English or Spanish will be excluded since these women are not eligible for the DA.
* history of invasive breast cancer
* Women with history ductal carcinoma in situ treated with radiation (since these women are generally not be eligible for radiation treatment)
* Paget's disease
* Inflammatory breast cancer
* A phyllodes tumor.
* In hospice
* Surgeon not willing to participate
* Psychiatric illness situations that would limit compliance with study requirements
* History of dementia
* Incapacity for informed consent
* Surgeon not willing to have patient complete study surveys
* 19 patients already successfully recruited that month and the patient is non-Hispanic white.

Primary Caregiver Exclusion Criteria:

* Age <18
* Non-English and non-Spanish speaking
* Psychiatric illness situations that would limit compliance with study requirements

Allied health professionals (Aim 4 at the end of the trial) Exclusion Criteria:

* A trainee
* Psychiatric illness situations that would limit compliance with study requirements

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 402 (Estimated)
Dates: Start 2026-02-04 (Estimated); Primary Completion 2032-10-01 (Estimated); Study Completion 2033-09-30 (Estimated)

PRIMARY OUTCOMES:
Receipt of aggressive treatment within 6 months of First Surgical Encounter (Arm A) | 6 months
  Research staff will review the medical records for all participants with eligible tumor and study characteristics seen by a participating surgeon during the trial to learn whether aggressive treatments were received (mastectomy, radiation treatment, sentinel lymph node biopsy [SLNB] or axillary dissections and/or systemic therapy) within 6 months of each participant's first surgical consultation.
Receipt of aggressive treatment within 6 months of First Surgical Encounter (Arm D) | 6 months
  Research staff will review the medical records for all participants with eligible tumor and study characteristics seen by a participating surgeon during the trial to learn whether aggressive treatments were received (mastectomy, radiation treatment, sentinel lymph node biopsy [SLNB] or axillary dissections and/or systemic therapy) within 6 months of each participant's first surgical consultation.

SECONDARY OUTCOMES:
Participant Perceived Shared Decision Making Quality Scale Score (Arm A) | at 1 week and at 6 months
  Assessed by the SDM Process Scale: 4 items-scored 0-4 with a total scores range of 0 to 16; patient/caregiver participant perspectives on how much surgeon reviewed reasons for having/not having radiotherapy after breast conserving surgery and for having SLNB. It also assesses if participants perceive being given a choice or asked about preferences.
Participant Perceived Shared Decision Making Quality Scale Score (Arm D) | at 1 week and at 6 months
  Assessed by the SDM Process Scale: 4 items-scored 0-4 with a total scores range of 0 to 16; patient/caregiver participant perspectives on how much surgeon reviewed reasons for having/not having radiotherapy after breast conserving surgery and for having SLNB. It also assesses if participants perceive being given a choice or asked about preferences.
Participant Decisional Conflict Scale Score (Arm A) | 1 week
  Assessed from patient/caregiver participants by the Decisional Conflict Scale of 10-items scored on three response options (0 "Yes," 4 "No," 2 "Unsure") for four subscales uncertainty, feeling informed, clear in one's values, and supported in the decision. A total scores range is 0 "No conflict" to 100 "extremely high conflict."
Participant Decisional Conflict Scale Score (Arm D) | 1 week
  Assessed from patient/caregiver participants by the Decisional Conflict Scale of 10-items scored on three response options (0 "Yes," 4 "No,"2 "Unsure") for four subscales assessing uncertainty, feeling informed, clear in one's values, and supported in the decision. A total scores range is 0 "No conflict" to 100 "extremely high conflict."
Participant Knowledge Score at 1 week (Arm A) | 1 week
  Assessed from patients/caregivers by 10 true/false items at 1 week about surgery and radiation. Total score is questions answered correctly (range 0-10)
Participant Knowledge Score at 6 Months (Arm A) | 6 months
  Assessed from patient/caregiver participants by 3 true/false items at 6 months about endocrine therapy. Total score is questions answered correctly (range 0-3).
Participant Knowledge Score at 1 week (Arm D) | 1 week
  Assessed patient/caregiver participants by 10 true/false items at 1 week about surgery and radiation. Total score is questions answered correctly (range 0-10)
Participant Knowledge Score at 6 Months (Arm D) | 6 months
  Assessed patient/caregiver participants by 3 true/false items at 6 months about endocrine therapy. Total score is questions answered correctly (range 0-3).
Subjective Financial Distress Index Score (Arm A) | 6 months
  Assessed by the Subjective Financial Distress index comprised of 14 items scored on three response options (0 "Not at All," 1 "Somewhat," and 2 "Very Much") with a scores range from 0-28. A higher score indicates higher financial toxicity.
Subjective Financial Distress Index Score (Arm D) | 6 months
  Assessed by the Subjective Financial Distress index comprised of 14 items scored on three response options (0 "Not at All," 1 "Somewhat," and 2 "Very Much") with a scores range from 0-28. A higher score indicates higher financial toxicity.
EuroQol EQ-5D-5L Scale Score (Arm A) | 1 week and 6 months
  Assessed by the 6-item EuroQol EQ-5D-5L descriptive system of 5 health dimensions that is scored on 5 response categories of "no problem/pain," "slight problems/pain," "moderate problems/pain," "severe problems/pain," and "unable/extreme pain/extremely anxious." The 5 responses give a health state or profile represented by a 5-digit number corresponding to response categories reported by participants for successive dimensions, beginning with mobility. Health states are scored to give the EQ-5D-5L index using a scoring algorithm from a value set derived from valuation tasks from general population samples.
EuroQol EQ-5D-5L Scale Score (Arm D) | 1 week and 6 months
  Assessed by the 6-item EuroQol EQ-5D-5L descriptive system of 5 health dimensions that is scored on 5 response categories of "no problem/pain," "slight problems/pain," "moderate problems/pain," "severe problems/pain," and "unable/extreme pain/extremely anxious." The 5 responses give a health state or profile represented by a 5-digit number corresponding to response categories reported by participants for successive dimensions, beginning with mobility. Health states are scored to give the EQ-5D-5L index using a scoring algorithm from a value set derived from valuation tasks from general population samples.
Change in Surgeon Self-Efficacy Scale Score from Baseline to End of Study (Arm B) | Baseline and at end of the study. End of study will vary from 6 months to 4 years
  Assessed by the Self-Efficacy Scale, surgeons report on 7 items scored on 7-point scale: 1 "strongly disagree" to 7 "strongly agree." A total score will be the mean and will range from 1 to 7. A higher score indicates greater self-efficacy.
Change in Surgeon Self-Efficacy Scale Score from Baseline to End of Study (Arm E) | Baseline and at end of the study. End of study will vary from 6 months to 4 years
  Assessed by the Self-Efficacy Scale, surgeons report 7 items scored on 7-point scale: 1 "strongly disagree" to 7 "strongly agree." A total score will be the mean and will range from 1 to 7. A higher score indicates greater self-efficacy.

CONTACTS AND LOCATIONS:
Overall Officials: Mara Schonberg, MD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (6):
- United States (6):
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Lahey Hospital and Medical Center, Burlington, Massachusetts
  - Beth Israel Deaconess Hospital, Needham, Massachusetts
  - Dana-Farber/Brigham and Women's Cancer Center at South Shore Hospital, Weymouth, Massachusetts

IPD SHARING:
Plan to Share IPD: Yes
All deidentified study data will be made available as public use data to the research community via a Harvard Dataverse Repository. Users will be required to agree to terms that prohibit unlawful uses and intentional violations of privacy, and require attribution. Use of the data will be otherwise unrestricted and free of charge.
Supporting Information: Study Protocol, Analytic Code
Time Frame: Data can be shared no earlier than one year following the date of publication or one year after completion of the grant.
Access Criteria: All deidentified study data will be made available as public use data to the research community via a Harvard Dataverse Repository. Users will be required to agree to terms that prohibit unlawful uses and intentional violations of privacy, and require attribution. Use of the data will be otherwise unrestricted and free of charge.

REFERENCES:
- [Background] Holmes-Rovner M, Kroll J, Schmitt N, Rovner DR, Breer ML, Rothert ML, Padonu G, Talarczyk G. Patient satisfaction with health care decisions: the satisfaction with decision scale. Med Decis Making. 1996 Jan-Mar;16(1):58-64. doi: 10.1177/0272989X9601600114. PMID 8717600
- [Background] McNaughton CD, Cavanaugh KL, Kripalani S, Rothman RL, Wallston KA. Validation of a Short, 3-Item Version of the Subjective Numeracy Scale. Med Decis Making. 2015 Nov;35(8):932-6. doi: 10.1177/0272989X15581800. Epub 2015 Apr 15. PMID 25878195
- [Background] Degner LF, Kristjanson LJ, Bowman D, Sloan JA, Carriere KC, O'Neil J, Bilodeau B, Watson P, Mueller B. Information needs and decisional preferences in women with breast cancer. JAMA. 1997 May 14;277(18):1485-92. PMID 9145723
- [Background] Brehaut JC, O'Connor AM, Wood TJ, Hack TF, Siminoff L, Gordon E, Feldman-Stewart D. Validation of a decision regret scale. Med Decis Making. 2003 Jul-Aug;23(4):281-92. doi: 10.1177/0272989X03256005. PMID 12926578
- [Background] Garvelink MM, Boland L, Klein K, Nguyen DV, Menear M, Bekker HL, Eden KB, LeBlanc A, O'Connor AM, Stacey D, Legare F. Decisional Conflict Scale Use over 20 Years: The Anniversary Review. Med Decis Making. 2019 May;39(4):301-314. doi: 10.1177/0272989X19851345. Epub 2019 May 29. PMID 31142194
- [Background] Fowler FJ Jr, Sepucha KR, Stringfellow V, Valentine KD. Validation of the SDM Process Scale to Evaluate Shared Decision-Making at Clinical Sites. J Patient Exp. 2021 Nov 26;8:23743735211060811. doi: 10.1177/23743735211060811. eCollection 2021. PMID 34869847
- [Background] McCreight MS, Rabin BA, Glasgow RE, Ayele RA, Leonard CA, Gilmartin HM, Frank JW, Hess PL, Burke RE, Battaglia CT. Using the Practical, Robust Implementation and Sustainability Model (PRISM) to qualitatively assess multilevel contextual factors to help plan, implement, evaluate, and disseminate health services programs. Transl Behav Med. 2019 Nov 25;9(6):1002-1011. doi: 10.1093/tbm/ibz085. PMID 31170296
- [Background] Glasgow RE, Harden SM, Gaglio B, Rabin B, Smith ML, Porter GC, Ory MG, Estabrooks PA. RE-AIM Planning and Evaluation Framework: Adapting to New Science and Practice With a 20-Year Review. Front Public Health. 2019 Mar 29;7:64. doi: 10.3389/fpubh.2019.00064. eCollection 2019. PMID 30984733
- [Background] Wagner TH, Yoon J, Jacobs JC, So A, Kilbourne AM, Yu W, Goodrich DE. Estimating Costs of an Implementation Intervention. Med Decis Making. 2020 Nov;40(8):959-967. doi: 10.1177/0272989X20960455. Epub 2020 Oct 20. PMID 33078681
- [Background] Falkenbach P, Raudasoja AJ, Vernooij RWM, Mustonen JMJ, Agarwal A, Aoki Y, Blanker MH, Cartwright R, Garcia-Perdomo HA, Kilpelainen TP, Lainiala O, Lamberg T, Nevalainen OPO, Raittio E, Richard PO, Violette PD, Tikkinen KAO, Sipila R, Turpeinen M, Komulainen J. Reporting of costs and economic impacts in randomized trials of de-implementation interventions for low-value care: a systematic scoping review. Implement Sci. 2023 Aug 21;18(1):36. doi: 10.1186/s13012-023-01290-3. PMID 37605243
- [Background] Schonberg MA, Jacobson AR, Karamourtopoulos M, Aliberti GM, Pinheiro A, Smith AK, Schuttner LC, Park ER, Hamel MB. Scripts and Strategies for Discussing Stopping Cancer Screening with Adults > 75 Years: a Qualitative Study. J Gen Intern Med. 2020 Jul;35(7):2076-2083. doi: 10.1007/s11606-020-05735-z. Epub 2020 Mar 3. PMID 32128689
- [Background] Jindal SK, Karamourtopoulos M, Jacobson AR, Pinheiro A, Smith AK, Hamel MB, Schonberg MA. Strategies for discussing long-term prognosis when deciding on cancer screening for adults over age 75. J Am Geriatr Soc. 2022 Jun;70(6):1734-1744. doi: 10.1111/jgs.17723. Epub 2022 Feb 28. PMID 35225351
- [Background] Minami CA, Bryan AF, Freedman RA, Revette AC, Schonberg MA, King TA, Mittendorf EA. Assessment of Oncologists' Perspectives on Omission of Sentinel Lymph Node Biopsy in Women 70 Years and Older With Early-Stage Hormone Receptor-Positive Breast Cancer. JAMA Netw Open. 2022 Aug 1;5(8):e2228524. doi: 10.1001/jamanetworkopen.2022.28524. PMID 36001314
- [Background] Schonberg MA, Li V, Marcantonio ER, Davis RB, McCarthy EP. Predicting Mortality up to 14 Years Among Community-Dwelling Adults Aged 65 and Older. J Am Geriatr Soc. 2017 Jun;65(6):1310-1315. doi: 10.1111/jgs.14805. Epub 2017 Feb 21. PMID 28221669
- [Background] Dossett LA, Mott NM, Bredbeck BC, Wang T, Jobin CT, Hughes TM, Hawley ST, Zikmund-Fisher BJ. Using Tailored Messages to Target Overuse of Low-Value Breast Cancer Care in Older Women. J Surg Res. 2022 Feb;270:503-512. doi: 10.1016/j.jss.2021.10.005. Epub 2021 Nov 19. PMID 34801801
- [Background] Carleton N, Zou J, Fang Y, Koscumb SE, Shah OS, Chen F, Beriwal S, Diego EJ, Brufsky AM, Oesterreich S, Shapiro SD, Ferris R, Emens LA, Tseng G, Marroquin OC, Lee AV, McAuliffe PF. Outcomes After Sentinel Lymph Node Biopsy and Radiotherapy in Older Women With Early-Stage, Estrogen Receptor-Positive Breast Cancer. JAMA Netw Open. 2021 Apr 1;4(4):e216322. doi: 10.1001/jamanetworkopen.2021.6322. PMID 33856473
- [Background] Stacey D, Lewis KB, Smith M, Carley M, Volk R, Douglas EE, Pacheco-Brousseau L, Finderup J, Gunderson J, Barry MJ, Bennett CL, Bravo P, Steffensen K, Gogovor A, Graham ID, Kelly SE, Legare F, Sondergaard H, Thomson R, Trenaman L, Trevena L. Decision aids for people facing health treatment or screening decisions. Cochrane Database Syst Rev. 2024 Jan 29;1(1):CD001431. doi: 10.1002/14651858.CD001431.pub6. PMID 38284415
- [Background] Schonberg MA, Birdwell RL, Bychkovsky BL, Hintz L, Fein-Zachary V, Wertheimer MD, Silliman RA. Older women's experience with breast cancer treatment decisions. Breast Cancer Res Treat. 2014 May;145(1):211-23. doi: 10.1007/s10549-014-2921-y. Epub 2014 Mar 31. PMID 24682710
- [Background] Chagpar AB, Horowitz N, Sanft T, Wilson LD, Silber A, Killelea B, Moran MS, DiGiovanna MP, Hofstatter E, Chung G, Pusztai L, Lannin DR. Does lymph node status influence adjuvant therapy decision-making in women 70 years of age or older with clinically node negative hormone receptor positive breast cancer? Am J Surg. 2017 Dec;214(6):1082-1088. doi: 10.1016/j.amjsurg.2017.07.036. Epub 2017 Sep 18. PMID 28939252
- [Background] Boughey JC, Haffty BG, Habermann EB, Hoskin TL, Goetz MP. Has the Time Come to Stop Surgical Staging of the Axilla for All Women Age 70 Years or Older with Hormone Receptor-Positive Breast Cancer? Ann Surg Oncol. 2017 Mar;24(3):614-617. doi: 10.1245/s10434-016-5740-z. Epub 2017 Jan 4. No abstract available. PMID 28054190
- [Background] Biganzoli L, Battisti NML, Wildiers H, McCartney A, Colloca G, Kunkler IH, Cardoso MJ, Cheung KL, de Glas NA, Trimboli RM, Korc-Grodzicki B, Soto-Perez-de-Celis E, Ponti A, Tsang J, Marotti L, Benn K, Aapro MS, Brain EGC. Updated recommendations regarding the management of older patients with breast cancer: a joint paper from the European Society of Breast Cancer Specialists (EUSOMA) and the International Society of Geriatric Oncology (SIOG). Lancet Oncol. 2021 Jul;22(7):e327-e340. doi: 10.1016/S1470-2045(20)30741-5. Epub 2021 May 14. PMID 34000244
- [Background] Liang S, Hallet J, Simpson JS, Tricco AC, Scheer AS. Omission of axillary staging in elderly patients with early stage breast cancer impacts regional control but not survival: A systematic review and meta-analysis. J Geriatr Oncol. 2017 Mar;8(2):140-147. doi: 10.1016/j.jgo.2016.12.003. Epub 2016 Dec 13. PMID 27986500
- [Background] Gentilini OD, Botteri E, Sangalli C, Galimberti V, Porpiglia M, Agresti R, Luini A, Viale G, Cassano E, Peradze N, Toesca A, Massari G, Sacchini V, Munzone E, Leonardi MC, Cattadori F, Di Micco R, Esposito E, Sgarella A, Cattaneo S, Busani M, Dessena M, Bianchi A, Cretella E, Ripoll Orts F, Mueller M, Tinterri C, Chahuan Manzur BJ, Benedetto C, Veronesi P; SOUND Trial Group. Sentinel Lymph Node Biopsy vs No Axillary Surgery in Patients With Small Breast Cancer and Negative Results on Ultrasonography of Axillary Lymph Nodes: The SOUND Randomized Clinical Trial. JAMA Oncol. 2023 Nov 1;9(11):1557-1564. doi: 10.1001/jamaoncol.2023.3759. PMID 37733364
- [Background] International Breast Cancer Study Group; Rudenstam CM, Zahrieh D, Forbes JF, Crivellari D, Holmberg SB, Rey P, Dent D, Campbell I, Bernhard J, Price KN, Castiglione-Gertsch M, Goldhirsch A, Gelber RD, Coates AS. Randomized trial comparing axillary clearance versus no axillary clearance in older patients with breast cancer: first results of International Breast Cancer Study Group Trial 10-93. J Clin Oncol. 2006 Jan 20;24(3):337-44. doi: 10.1200/JCO.2005.01.5784. Epub 2005 Dec 12. PMID 16344321
- [Background] Martelli G, Boracchi P, Ardoino I, Lozza L, Bohm S, Vetrella G, Agresti R. Axillary dissection versus no axillary dissection in older patients with T1N0 breast cancer: 15-year results of a randomized controlled trial. Ann Surg. 2012 Dec;256(6):920-4. doi: 10.1097/SLA.0b013e31827660a8. PMID 23154393
- [Background] Mann GB, Skandarajah AR, Zdenkowski N, Hughes J, Park A, Petrie D, Saxby K, Grimmond SM, Murugasu A, Spillane AJ, Chua BH, Badger H, Braggett H, Gebski V, Mou A, Collins JP, Rose AK. Postoperative radiotherapy omission in selected patients with early breast cancer following preoperative breast MRI (PROSPECT): primary results of a prospective two-arm study. Lancet. 2024 Jan 20;403(10423):261-270. doi: 10.1016/S0140-6736(23)02476-5. Epub 2023 Dec 5. PMID 38065194
- [Background] Potter R, Gnant M, Kwasny W, Tausch C, Handl-Zeller L, Pakisch B, Taucher S, Hammer J, Luschin-Ebengreuth G, Schmid M, Sedlmayer F, Stierer M, Reiner G, Kapp K, Hofbauer F, Rottenfusser A, Postlberger S, Haider K, Draxler W, Jakesz R; Austrian Breast and Colorectal Cancer Study Group. Lumpectomy plus tamoxifen or anastrozole with or without whole breast irradiation in women with favorable early breast cancer. Int J Radiat Oncol Biol Phys. 2007 Jun 1;68(2):334-40. doi: 10.1016/j.ijrobp.2006.12.045. Epub 2007 Mar 23. PMID 17363187
- [Background] Kunkler IH, Williams LJ, Jack WJL, Cameron DA, Dixon JM. Breast-Conserving Surgery with or without Irradiation in Early Breast Cancer. N Engl J Med. 2023 Feb 16;388(7):585-594. doi: 10.1056/NEJMoa2207586. PMID 36791159
- [Background] Kunkler IH, Williams LJ, Jack WJ, Cameron DA, Dixon JM; PRIME II investigators. Breast-conserving surgery with or without irradiation in women aged 65 years or older with early breast cancer (PRIME II): a randomised controlled trial. Lancet Oncol. 2015 Mar;16(3):266-73. doi: 10.1016/S1470-2045(14)71221-5. Epub 2015 Jan 28. PMID 25637340
- [Background] Chesney TR, Yin JX, Rajaee N, Tricco AC, Fyles AW, Acuna SA, Scheer AS. Tamoxifen with radiotherapy compared with Tamoxifen alone in elderly women with early-stage breast cancer treated with breast conserving surgery: A systematic review and meta-analysis. Radiother Oncol. 2017 Apr;123(1):1-9. doi: 10.1016/j.radonc.2017.02.019. PMID 28391871
- [Background] Gennari R, Curigliano G, Rotmensz N, Robertson C, Colleoni M, Zurrida S, Nole F, de Braud F, Orlando L, Leonardi MC, Galimberti V, Intra M, Veronesi P, Renne G, Cinieri S, Audisio RA, Luini A, Orecchia R, Viale G, Goldhirsch A. Breast carcinoma in elderly women: features of disease presentation, choice of local and systemic treatments compared with younger postmenopasual patients. Cancer. 2004 Sep 15;101(6):1302-10. doi: 10.1002/cncr.20535. PMID 15316944
- [Background] Schonberg MA, Karamourtopoulos M, Jacobson AR, Aliberti GM, Pinheiro A, Smith AK, Davis RB, Schuttner LC, Hamel MB. A Strategy to Prepare Primary Care Clinicians for Discussing Stopping Cancer Screening With Adults Older Than 75 Years. Innov Aging. 2020 Jul 7;4(4):igaa027. doi: 10.1093/geroni/igaa027. eCollection 2020. PMID 32793815
- [Background] Schonberg MA, Freedman RA, Recht AR, Jacobson AR, Aliberti GM, Karamourtopoulos M, Nakhlis F, McCarthy EP, Pories SE, Sharma R, Dominici LS. Developing a patient decision aid for women aged 70 and older with early stage, estrogen receptor positive, HER2 negative, breast cancer. J Geriatr Oncol. 2019 Nov;10(6):980-986. doi: 10.1016/j.jgo.2019.05.004. Epub 2019 May 24. PMID 31130442
- [Background] Minami CA, Freedman RA, Karamourtopoulos M, Pinheiro A, Gilliam E, Aliberti G, Pories SE, Recht A, Lotz M, Dominici LS, Schonberg MA. Acceptability of a patient decision aid for women aged 70 and older with stage I, estrogen receptor-positive, HER2-negative breast cancer. J Geriatr Oncol. 2021 Jun;12(5):724-730. doi: 10.1016/j.jgo.2021.02.028. Epub 2021 Mar 5. PMID 33678596
- [Background] Fyles AW, McCready DR, Manchul LA, Trudeau ME, Merante P, Pintilie M, Weir LM, Olivotto IA. Tamoxifen with or without breast irradiation in women 50 years of age or older with early breast cancer. N Engl J Med. 2004 Sep 2;351(10):963-70. doi: 10.1056/NEJMoa040595. PMID 15342804
- [Background] Sarkar U, Schillinger D, Lopez A, Sudore R. Validation of self-reported health literacy questions among diverse English and Spanish-speaking populations. J Gen Intern Med. 2011 Mar;26(3):265-71. doi: 10.1007/s11606-010-1552-1. Epub 2010 Nov 6. PMID 21057882
- [Background] Bychkovsky BL, Schonberg MA. Poor persistence with hormonal therapy among women with breast cancer. J Geriatr Oncol. 2016 May;7(3):154-7. doi: 10.1016/j.jgo.2016.04.002. Epub 2016 Apr 28. No abstract available. PMID 27133286
- [Background] Lee SJ, Leipzig RM, Walter LC. Incorporating lag time to benefit into prevention decisions for older adults. JAMA. 2013 Dec 25;310(24):2609-10. doi: 10.1001/jama.2013.282612. No abstract available. PMID 24322396
- [Background] Glasgow RE, Vogt TM, Boles SM. Evaluating the public health impact of health promotion interventions: the RE-AIM framework. Am J Public Health. 1999 Sep;89(9):1322-7. doi: 10.2105/ajph.89.9.1322. PMID 10474547
- [Background] Shickh S, Leventakos K, Lewis MA, Bombard Y, Montori VM. Shared Decision Making in the Care of Patients With Cancer. Am Soc Clin Oncol Educ Book. 2023 Jun;43:e389516. doi: 10.1200/EDBK_389516. PMID 37339391
- [Background] Tseng J, Bazan JG, Minami CA, Schonberg MA. Not Too Little, Not Too Much: Optimizing More Versus Less Locoregional Treatment for Older Patients With Breast Cancer. Am Soc Clin Oncol Educ Book. 2023 Jun;43:e390450. doi: 10.1200/EDBK_390450. PMID 37327467
- [Background] Hawkins AT, Fayanju OM, Maduekwe UN. Shared Decision-Making in the Surgical Sciences. JAMA Surg. 2023 Nov 1;158(11):1121-1122. doi: 10.1001/jamasurg.2023.2396. PMID 37466987
- [Background] Simmons L, Leavitt L, Ray A, Fosburgh B, Sepucha K. Shared Decision Making in Common Chronic Conditions: Impact of a Resident Training Workshop. Teach Learn Med. 2016;28(2):202-9. doi: 10.1080/10401334.2016.1146600. PMID 27064722
- [Background] Sepucha KR, Simmons LH, Barry MJ, Edgman-Levitan S, Licurse AM, Chaguturu SK. Ten Years, Forty Decision Aids, And Thousands Of Patient Uses: Shared Decision Making At Massachusetts General Hospital. Health Aff (Millwood). 2016 Apr;35(4):630-6. doi: 10.1377/hlthaff.2015.1376. PMID 27044963
- [Background] Stacey D, Samant R, Bennett C. Decision making in oncology: a review of patient decision aids to support patient participation. CA Cancer J Clin. 2008 Sep-Oct;58(5):293-304. doi: 10.3322/CA.2008.0006. Epub 2008 Aug 28. PMID 18755939
- [Background] Hind D, Wyld L, Beverley CB, Reed MW. Surgery versus primary endocrine therapy for operable primary breast cancer in elderly women (70 years plus). Cochrane Database Syst Rev. 2006 Jan 25;(1):CD004272. doi: 10.1002/14651858.CD004272.pub2. PMID 16437480
- [Background] Holmes-Rovner M. International Patient Decision Aid Standards (IPDAS): beyond decision aids to usual design of patient education materials. Health Expect. 2007 Jun;10(2):103-7. doi: 10.1111/j.1369-7625.2007.00445.x. No abstract available. PMID 17524003
- [Background] Minami CA, Jin G, Freedman RA, Schonberg MA, King TA, Mittendorf EA. Trends in Locoregional Therapy in Older Women with Early-Stage Hormone Receptor-Positive Breast Cancer by Frailty and Life Expectancy. Ann Surg Oncol. 2024 Feb;31(2):920-930. doi: 10.1245/s10434-023-14446-8. Epub 2023 Oct 18. PMID 37851196
- [Background] Schonberg MA, Marcantonio ER, Ngo L, Silliman RA, McCarthy EP. Does Life Expectancy Affect Treatment of Women Aged 80 and Older with Early Stage Breast Cancers? J Geriatr Oncol. 2012 Jan 1;3(1):8-16. doi: 10.1016/j.jgo.2011.10.002. PMID 22368726
- [Background] Diab SG, Elledge RM, Clark GM. Tumor characteristics and clinical outcome of elderly women with breast cancer. J Natl Cancer Inst. 2000 Apr 5;92(7):550-6. doi: 10.1093/jnci/92.7.550. PMID 10749910
- [Background] Schonberg MA, Marcantonio ER, Li D, Silliman RA, Ngo L, McCarthy EP. Breast cancer among the oldest old: tumor characteristics, treatment choices, and survival. J Clin Oncol. 2010 Apr 20;28(12):2038-45. doi: 10.1200/JCO.2009.25.9796. Epub 2010 Mar 22. PMID 20308658